CLINICAL TRIAL: NCT07264972
Title: Constitution d'Une Collection Biologique à Des Fins de Recherche médicale Pour Les Patients du Centre de référence Des Maladies Rares Des Vaisseaux du Cerveau et de l'Oeil à l'hôpital Lariboisière
Brief Title: Creation of a Biological Collection for Medical Research Purposes for Patients at the Reference Center for Rare Diseases of the Blood Vessels of the Brain and Eye at Lariboisière Hospital
Acronym: B-MRVC
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200773
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cerebrovascular Disease
Keywords: rare cerebrovascular disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients with rare cerebrovascular disease
  Interventions: Other: additional samples for research purposes

INTERVENTIONS:
Other: additional samples for research purposes — Blood and urine sampling

SUMMARY:
The aim of establishing a biological collection associated with the existing rare cerebral vascular disease cohort is to identify new prognostic or disease progression biomarkers that could improve patient care or identify new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a rare cerebral vascular disease of the brain, including:

Familial intracranial aneurysms, cerebral amyloid angiopathy, CADASIL, familial cerebral cavernoma, familial cervical or intracranial artery dissection, vascular leukoencephalopathy (hereditary), familial hemiplegic migraine, cerebral arteriovenous malformation, moya-moya, cerebral venous thrombosis, hereditary retinal tortuosity, cerebro-retinal vasculopathies, other known rare diseases, or other rare diseases that are undetermined or not yet described.

* Participation in the MVCR cohort
* Adults >18 years old
* Affiliation with French social security or beneficiary - Signature of informed consent

Exclusion Criteria:

* Incompatibility with long-term follow-up at CERVCO
* Patient under guardianship/conservatorship
* Pregnant or breastfeeding women
* Patient under AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rare cerebrovascular diseases
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Time required for sample storage (freezing) to ensure the stability of most measurable elements in a biological sample | Up to 2 years after inclusion
  for each sample

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisière hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided